CLINICAL TRIAL: NCT04830670
Title: Comparison of Bone Formation According to Different Maxillary Sinus Width: a Multicenter Prospective Study.
Brief Title: Bone Formation Maxillary Sinus Width
Status: Completed | Type: Observational
Sponsor: International Piezosurgery Academy (Other)
Responsible Party: Sponsor
Other Study IDs: WIDE&NARROW
Record Dates: First submitted 2021-03-25; First posted 2021-04-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Alveolar Bone Resorption
Keywords: Sinus lift;; sinus elevation;; sinus width;; bone graft; histomorphometry; alveolar bone atrophy
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — alveolar bone specimen containing native bone, regenerated bone (with residual graft particles); the specimens were retrieved with a trephine bur that prepared the same time the implant site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Large sinus: same patient, sinus width > 12mm measured at 10mm from the alveolar crest at the planned implant site
  Interventions: Procedure: sinus floor elevation with lateral approach
- narrow sinus: same patient, sinus width < 12mm measured at 10mm from the alveolar crest at the planned implant site
  Interventions: Procedure: sinus floor elevation with lateral approach

INTERVENTIONS:
Procedure: sinus floor elevation with lateral approach — sinus floor elevation with lateral approach. 6 months healing phase. implant site preparation with trephine bur and bone specimen retrieval.

SUMMARY:
According to previous scientific evidence lining on biological concept of bone regeneration into the maxillary sinus, an observational study was set up to record possible (hypothesized) difference in bone formation between different width of the maxillary sinus itself. Therefore, a multicenter study was set up that foresaw a surgical intervention of sinus lift with lateral approach, the 6 months healing phase, the implant insertion in two sites with the implant site preparation made by a trephine bur to retrieve a bone specimen for histomorphometric examination without any additive invasively for the patient.

DETAILED DESCRIPTION:
Material and Methods Study protocol This study was designed as a multicenter prospective study following STROBE (STrengthening the Reporting of Observational studies in Epidemiology) guidelines. All procedures were performed in strict accordance with the recommendations of the Declaration of Helsinki as revised in Fortaleza for investigations with human subjects. The study protocol had been approved by the relevant ethical committee (Comitato Etico Calabria-Sezione Area Nord n. 55/2016). Patients, after being thoroughly informed about the study protocol, the treatment, its alternatives and any potential risk, signed a written informed consent for the participation in the study and authorized the use of their data for research purposes.

Any patient with Kennedy class II partial edentulism requiring unilateral sinus floor elevation for the placement of two not adjacent dental implants supporting a fixed partial prosthesis was eligible for entering this study.

Pre-surgical phase Patients recruited in the present study underwent a careful clinical examination, including assessment of periodontal conditions (probing and periapical radiographs), evaluation of available bone volume in the edentulous areas on cone beam computed tomography and analysis of occlusal relationships (diagnostic wax-up). A surgical resin guide was manufactured by duplicating the diagnostic wax-up.

All patients received professional mechanical tooth cleaning and periodontal debridement one week prior to surgery and were prescribed with chlorhexidine digluconate 0.2% mouthwash twice a day.

Surgical procedure All patients underwent antibiotic prophylaxis (2 g single-dose amoxicillin one hour before surgery). After performing local anaesthesia (articaine 4% with epinephrine 1:100.000) and elevating a full-thickness flap, the surgical guide was placed in position and an antrostomy was created by consuming the lateral wall of the maxillary sinus with ultrasonic instrumentation in the area between the two planned implant sites. The sinus membrane was then carefully elevated and, after checking its integrity with visual inspection and Valsalva maneuver, the subantral space was filled with a composite graft in granules [50% cortico-cancellous porcine graft (Gen-Os, Tecnoss, Pianezza, Italy) - 50% synthetic nano-hydroxyapatite (Fisiograft Bone, Ghimas, Casalecchio di Reno, Italy)]. A resorbable bovine collagen membrane (Bio-Gide, Geistlich, Wolhusen, Switzerland) fixed with two pins was placed to cover the lateral antrostomy and flaps were sutured with Sentineri sutures and single stitches using synthetic monofilament. Patients were prescribed with antibiotics for 4 days (amoxicillin 1 g three times a day) and NSAID (ibuprofen 600 mg), when needed. Sutures were removed after 10 days.

After 6 months of healing, a cone beam tc scan was performed to evaluate the radiographic outcome of the regenerative procedure and to plan implant insertion. With the assistance of the surgical template, two bone-core biopsy biopsies were harvested in the planned implant sites by using 3-mm diameter trephine drills (2982.Y0.30, DenTag, Maniago, Italy) (Fig. 3-4). Dental implants were then inserted in the biopsy sites: after 5 months of submerged healing, they were restored with screwed ceramic crowns.

Radiographic measurements Radiographic measurements were taken from the three cone beam CT cross-sectional slices (step 1 mm; width 1 mm) corresponding to the position where the biopsy was retrieved. Two independent calibrated examiners (A.R. and Fe.Be.) measured residual bone height (RBH) between the alveolar ridge and the sinus floor; sinus width (SW) (distance between buccal and palatal walls at 10-mm level, comprising the residual alveolar crest. Distances were measured by using the specific tool of an imaging software (OsiriX MD, Pixmeo SARL, Bernex, Switzerland) and were expressed in millimeters. Intra-examiner reliability was assessed with Cohen's K test.

Sample processing for histological analysis Histologic and histomorphometric analyses of all specimens were performed by one of the authors (VN), blinded to the study design and to biopsy origin. Immediately after harvesting, biopsies were carefully rinsed with cold 5% glucose solution to remove blood remnants maintaining the correct osmolarity (278 milliosmole/L).

Specimens were subsequently fixed for three days in 10% buffered formalin solution at pH 7.2, and then dehydrated in an ascending series of alcohol rinses and embedded in a methacrylate resin (Technovit 7200 VLC, Kulzer, Wehrheim, Germany). After 12 days of polymerization, biopsies were cut along their longitudinal axis with a high-precision carborundum disk at 50 µm and then ground down under running water with a series of polishing discs to about 30 ± 10 µm. The slides were then mounted and stained with acid fuchsine-toluidine blue and von Kossa staining.

Histomorphometry The following variables were measured for each biopsy: total area of the biopsy (in mm2), percentage of newly-formed bone (NFB),percentage of connective tissue/marrow spaces (MS), and percentage of residual graft particles (RG). The analysis was performed using transmitted brightfield light microscope (Biostar B3; Exacta Optech, San Prospero, Italy), connected to high resolution digital camera (Moticam 5.0; Motic Microscopy, Kowloon, China). A software with image capturing capabilities (Image-Pro Plus 6.0; Media Cybernetics Inc., Bethesda, MD, U.S.A.) was used to analyze images. Software calibration was performed for each image analysis by using the "Calibration Wizard" tool, which reports the number of pixels between two selected points. Linear remapping of the pixel numbers was used to calibrate the distance in µm or in mm according to the magnification degree.

Predictor and outcome variables This prospective study tested the null hypothesis of no differences in new bone formation among areas of different width in the same sinus against the alternative hypothesis of a difference.

The primary predictor variables were sinus width (SW) and residual bone height (RBH).

Primary outcome measure:

• new bone formation (NFB) after six months of healing

Secondary outcome measures:

* residual graft (RG): after six months of healing
* any complications or adverse events

Sample size calculation and statistical power A statistical software (Statistica per Discipline Biomediche, Version 6.0, Mc Graw-Hill, New York, NY, U.S.A.) was used to determine the sample size of this prospective study, basing on data of a previous publication. Expected difference in NFB (as mean percentage) between narrow and wide part of the sinus was 13.8±18.25% (using sinus width=13 mm as a cut-off). A sample of 16 histological specimens for each group was required to detect significant differences between the two groups (confidence level 5% with statistical power of 80%).

Statistical analysis An independent investigator (A.R.) analyzed all datasets with statistical software (IBM SPSS Statistics for Windows, Version 25.0, IBM Corp., Armonk, NY, USA). Data normality was assessed with Shapiro-Wilk test: all datasets met the required assumptions for using parametric methods. Descriptive statistics included mean and standard deviation. The value of α was set to 0.05.

Differences in NFB between mesial and distal sites were evaluated by means of paired samples t-test. The potential influence of sinus width and RBH on NFB and RG percentage was evaluated by using Pearson correlation coefficient.

ELIGIBILITY:
Inclusion Criteria:

* height of the residual bone crest <5 mm in both sites where implant placement was planned;
* age >18 years;
* written informed consent given.

Exclusion Criteria:

* general contraindications to implant surgery
* smokers
* uncontrolled diabetes (HBA1c > 7.5%)
* treated or under treatment with intravenous antiresorptive drugs
* allergy to bovine collagen
* immunosuppressed
* irradiated in the head and neck area
* pregnant or breastfeeding
* substance abusers
* psychiatric problems or unrealistic expectations
* patient not fully able to comply with the study protocol.
* maxillary sinus conditions contraindicating sinus floor elevation
* poor oral hygiene and motivation (FMPS >25 and or FMBS>20)
* Schneiderian membrane perforation during surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any patient with Kennedy class II partial edentulism (Kennedy 1928) requiring unilateral sinus floor elevation for the placement of two not adjacent dental implants supporting a fixed partial prosthesis was eligible for entering this study
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
quantity (%) of newly formed bone | 6 months
  quantity (%) of newly formed bone (NFB) in histomorphometric analysis

SECONDARY OUTCOMES:
quantity (%) of graft | 6 months
  quantity (%) of residual graft (RG) in histomorphometric analysis
quantity of complications | through study completion, an average of 1 year
  quantity of any complications or adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Stacchi, Dr., Principal Investigator — Piezoelectricsurgery Academy
Locations (3):
- Italy (3):
  - Hesire, Cassano Allo Ionio, CS
  - Studio, Gorizia, GO
  - Studio B, Verona, VR

IPD SHARING:
Plan to Share IPD: No
data will be shared after data managing and statistics

REFERENCES:
- [Result] Stacchi C, Spinato S, Lombardi T, Bernardello F, Bertoldi C, Zaffe D, Nevins M. Minimally Invasive Management of Implant-Supported Rehabilitation in the Posterior Maxilla, Part I. Sinus Floor Elevation: Biologic Principles and Materials. Int J Periodontics Restorative Dent. 2020 May/Jun;40(3):e85-e93. doi: 10.11607/prd.4497. PMID 32233183
- [Result] Stacchi C, Spinato S, Lombardi T, Bernardello F, Bertoldi C, Zaffe D, Nevins M. Minimally Invasive Management of Implant-Supported Rehabilitation in the Posterior Maxilla, Part II. Surgical Techniques and Decision Tree. Int J Periodontics Restorative Dent. 2020 May/Jun;40(3):e95-e102. doi: 10.11607/prd.4498. PMID 32233185
- [Result] Stacchi C, Vercellotti T, Toschetti A, Speroni S, Salgarello S, Di Lenarda R. Intraoperative complications during sinus floor elevation using two different ultrasonic approaches: a two-center, randomized, controlled clinical trial. Clin Implant Dent Relat Res. 2015 Jan;17 Suppl 1:e117-25. doi: 10.1111/cid.12136. Epub 2013 Aug 22. PMID 23968289
- [Result] Avila G, Wang HL, Galindo-Moreno P, Misch CE, Bagramian RA, Rudek I, Benavides E, Moreno-Riestra I, Braun T, Neiva R. The influence of the bucco-palatal distance on sinus augmentation outcomes. J Periodontol. 2010 Jul;81(7):1041-50. doi: 10.1902/jop.2010.090686. PMID 20450402